CLINICAL TRIAL: NCT04202796
Title: Catheter Ablation in Congenital Heart Disease: French National Prospective Registry
Acronym: CATCH-Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paris Cardiovascular Research Center (Inserm U970) (Other Government)
Collaborators: European Georges Pompidou Hospital (Other); Centre Chirurgical Marie Lannelongue (Other); Clinique Pasteur Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: MR2C2001
Record Dates: First submitted 2019-12-15; First posted 2019-12-18 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Congenital Heart Disease; Arrhythmia
Keywords: catheter ablation
MeSH Terms: conditions — Heart Defects, Congenital; Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Catheter ablation — Catheter ablation of arrhythmia

SUMMARY:
Arrhythmias represent one of the main late complications in patients with congenital heart disease. Atrial arrhythmias are associated with a significant morbidity and are the first cause of urgent hospitalization, and sudden death from ventricular arrhythmias is a leading cause of death in this population.

The exponential increase of the number of patients with congenital heart disease and the improvement of ablative technologies are associated with a significant increase of the number of catheter ablation procedures.

Most of available studies are retrospective or include a limited number of patients.

The aim of this study is to assess the efficacy of catheter ablation in patients with congenital heart disease through a national prospective registry. Secondary objectives are i) to identify factors associated with catheter ablation efficacy in different cardiac defects, ii) to describe complications associated with catheter ablation in this specific population, and iii) to assess the impact of catheter ablation on quality of life of patients with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients with congenital heart disease referred for catheter ablation

Exclusion Criteria:

* Absence of patient's consent
* Patient under guardianship or curatorship
* Pregnant woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with congenital heart disease referred for catheter ablation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of targeted arrhythmia | 12 months
  Rate of freedom from targeted arrhythmia recurrence

SECONDARY OUTCOMES:
Recurrence of any arrhythmia | 12 months
  Rate of freedom from any arrhythmia recurrence at 12 months
Long-term recurrence of targeted and any arrhythmia | 24 months
  Rate of freedom from targeted and any arrhythmia recurrence
Complications | 1 month
  Complications associated with catheter ablation
Quality of life assessed by SF36 score | 6 months
  Quality of life change before and after catheter ablation assessed by SF36 score
Quality of life assessed by EQ5D3L score | 6 months
  Quality of life change before and after catheter ablation assessed by EQ5D3L score

CONTACTS AND LOCATIONS:
Overall Officials: Victor Waldmann, MD, MPH, Principal Investigator — Paris Cardiovascular Research Center (Inserm U970)
Locations (1):
- Georges Pompidou European Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No